CLINICAL TRIAL: NCT00624559
Title: COX-2 Regulation of Renal Sodium Handling in Blood Pressure Maintenance
Brief Title: The Role of COX-2 Inhibition in Salt Sensitivity of Blood Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, William Farquhar, Associate Professor and Department Chair, KAAP, University of Delaware
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 134024-1
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Results first posted 2011-12-21 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension
Keywords: Salt sensitivity of Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Celebrex; Low sodium (Experimental): Subject completes a normal sodium diet (3 days), a low salt diet (7 days), followed by a high salt diet (7 days) while taking a celebrex pill (100 mg twice a day for 17 day trial), randomized for trial order (drug versus placebo) and sodium diet order (low versus high sodium).
  Interventions: Drug: celecoxib (Celebrex)
- Celebrex, High Sodium (Experimental): Subject completes a normal sodium diet (3 days), a high salt diet (7 days), followed by a low salt diet (7 days) while taking a celebrex pill (100 mg twice a day for 17 day trial), randomized for trial order (drug versus placebo) and sodium diet order (low versus high sodium).
  Interventions: Drug: celecoxib (Celebrex)
- Placebo, Low Sodium (Placebo Comparator): Subject completes a normal sodium diet (3 days), a low salt diet (7 days), followed by a high salt diet (7 days) while taking a placebo pill (twice a day for 17 day trial), randomized for trial order (drug versus placebo) and sodium diet order (low versus high sodium).
  Interventions: Other: Placebo
- Placebo, High Sodium (Placebo Comparator): Subject completes a normal sodium diet (3 days), a high salt diet (7 days), followed by a low salt diet (7 days) while taking a placebo pill (twice a day for 17 day trial), randomized for trial order (drug versus placebo) and sodium diet order (low versus high sodium).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: celecoxib (Celebrex) — Celecoxib (Celebrex) was administered at 100 mg, twice per day for each day of sodium diet
  Other Names: Celebrex
  Arms: Celebrex, High Sodium; Celebrex; Low sodium
Other: Placebo — Placebo pill taken twice per day on each day of the diet
  Arms: Placebo, High Sodium; Placebo, Low Sodium

SUMMARY:
The purpose of this study is to determine if the drug Celebrex changes the way the kidney gets rid of salt and maintains blood pressure.

DETAILED DESCRIPTION:
There have been many studies done with analgesics such as acetaminophen and non-steroidal anti-inflammatory drugs; however it is not understood how blood pressure changes while using Celebrex. The study hypothesis is that Celebrex will increase salt sensitivity of blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women

Exclusion Criteria:

* history of heart disease
* have had heart surgery
* high blood pressure
* diabetes
* cancer
* any other disease such as kidney or neurological diseases
* taking medications such as aspirin or medicines for your heart or blood pressure
* have asthma or are allergic to sulfa drugs
* body mass index greater than 30
* use tobacco
* pregnant
* women using oral contraceptives or hormone replacement therapy

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Farquhar, PhD, Principal Investigator — University of Delaware; Michael Stillabower, MD, Study Director — Christiana Care Health Services
Locations (1):
- University of Delaware, Newark, Delaware, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Celebrex, High Sodium: Each subject completes a normal sodium diet (3 days), a high salt diet (7 days), and a low salt diet (7 days) while taking either a placebo or celebrex (each trial is 17 days long). Each subject completes 2 full 17 day trials (one month 'washout' between each trial); one time taking the placebo and one taking celebrex (randomized).
- Celebrex, Low Sodium: 100 mg Celebrex, twice per day for 7 days on low sodium diet
- Placebo, Low Sodium; Placebo, High Sodium: Placebo pill taken twice per day over the course of the diet
Period: Overall Study
Arm/Group | Celebrex, High Sodium | Celebrex, Low Sodium | Placebo, Low Sodium | Placebo, High Sodium
Started | 3 (Celebrex 1st: 3days baseline(100mmol), 7days high(350mmol) followed by 7days low(20mmol) sodium/day) | 3 (Celebrex 1st: 3days baseline(100mmol), 7days low(20mmol) followed by 7days high(350mmol) sodium/day) | 3 (Placebo 1st: 3days baseline(100mmol), 7days low(20mmol) followed by 7days high(350mmol) sodium/day) | 3 (Placebo 1st: 3days baseline(100mmol), 7days high(350mmol) followed by 7days low(20mmol) sodium/day)
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celebrex, High Sodium | Celebrex, Low Sodium | Placebo, Low Sodium | Placebo, High Sodium | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 3 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35 (2) | 35 (2) | 35 (2) | 35 (2) | 35 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 2
  Male | 3 | 2 | 2 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Pressure
Description: Blood pressure was measured on the last day of each 7 day sodium diet for 24 hours using an ambulatory blood pressure monitor
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Celebrex, Low Sodium Diet: Result taken at the end of 7 day low sodium diet
- Celebrex, High Sodium Diet: Result taken on last day of a 7 day high salt diet
- Placebo, Low Sodium Diet: Blood pressure taken over 24 hours on the last day of the low sodium diet with and ambulatory blood pressure monitor
- Placebo, High Sodium Diet: Blood pressure taken with an ambulatory blood pressure monitor, over 24 hours on the last day of the high sodium diet
Arm/Group | Celebrex, Low Sodium Diet | Celebrex, High Sodium Diet | Placebo, Low Sodium Diet | Placebo, High Sodium Diet
Number analyzed (Participants) | 12 | 12 | 12 | 12
mm Hg | 88 (2) | 87 (2) | 87 (2) | 87 (2)

2. Secondary Outcome: Urinary Sodium Excretion
Description: Urine collected over 24 hour period on last day of each different sodium diet
Time Frame: 24 hour
Measure: Mean (Standard Error); unit: mmol Na+/24 hr
Arm/Group | Celebrex, Low Sodium Diet | Celebrex, High Sodium Diet | Placebo, Low Sodium Diet | Placebo, High Sodium Diet
Number analyzed (Participants) | 12 | 12 | 12 | 12
mmol Na+/24 hr | 17 (7) | 281 (27) | 14 (3) | 253 (10)

ADVERSE EVENTS:
Arm/Group | Celebrex, High Sodium | Celebrex, Low Sodium | Placebo, Low Sodium | Placebo, High Sodium
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No